CLINICAL TRIAL: NCT02118090
Title: Assessing Chloroquine Resistance of Plasmodium Vivax in Malaria Endemic Area
Brief Title: Assessment of Plasmodium Vivax Chloroquine Resistance in Cambodia:
Acronym: CRePViCam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Pasteur, Cambodia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Didier Menard, Malaria Molecular Epidemiology Unit, Institut Pasteur, Cambodia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPC_Pv_CQR_RTK; R01AI103228 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Vivax Malaria
Keywords: malaria; Plasmodium vivax; drug resistance; chloroquine; Cambodia
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — Chloroquine; 2,6-diisopropylphenol docosahexaenoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine (Experimental): Patients treat with chloroquine sulfate (NIVAQUINE) 10 mg/kg/day - 3 days
  Interventions: Drug: Chloroquine sulfate
- DHA-PP (Active Comparator): Patient treat with DHA 40 mg and PP 320 mg, (Duo-Cotecxin®) The approximate total adult dose is 2-4 mg/kg for DHA and 20mg/kg for PP
  Interventions: Drug: DHA-PP

INTERVENTIONS:
Drug: Chloroquine sulfate — Chloroquine sulfate (NIVAQUINE) - 30 mg/kg for 3 days
  Other Names: NIVAQUINE
  Arms: Chloroquine
Drug: DHA-PP — DHA-PIP (Duo-Cotecxin®, DHA 40 mg and PP 320 mg, Zhejiang Holley Nanhu Pharamaceutical Co. Ltd, Jiaxing, Zhejiang province, China): one tablet of DHA-PIP contains 40 mg of dihydroartemisinin (DHA) and 320 mg piperaquine (PIP). It is an oral administration, one dose a day for 3 consecutive days. An adult dose (≥40 kg to 60kg body weight or more than 15 years old) consisted of three doses of 3 tablets over consecutive days (Total dose 9 tablets). The approximate total adult dose was 2-4 mg/kg for DHA and 20mg/kg for PP.
  Other Names: Duo-Cotecxin
  Arms: DHA-PP

SUMMARY:
The investigators propose to leverage the unique infrastructures and expertise of National Centre for Parasitology Entomology and Malaria Control and the Pasteur Institute in Cambodia and combine modern fieldwork, including a mobile laboratory fully equipped for molecular biology and culture experiments, with state-of-the-art genomic analyses to investigate how Plasmodium vivax parasites respond to antimalarial drugs. The investigators will focus on resistance to CQ, the choice treatment for vivax malaria in most endemic countries, for which treatment failures have been reported in Cambodia. The study will address some of the key biological mechanisms limiting the efficiency of drug therapy in P. vivax, including the identification of genetic polymorphisms underlying drug resistance in Cambodian P. vivax. The findings will provide a first unbiased perspective on the mechanisms of drug resistance in P. vivax and have the strong potential to significantly improve malaria control in Southeast Asia.

DETAILED DESCRIPTION:
In order to assess the resistance phenotype of P. vivax to CQ, the methodology will involve the following steps:

1. Inclusion of P.vivax mono-infected patients from villages in treatment failure-reported area (Ban Lung district, Rattanakiri)
2. Pv diagnostic confirmation (microscopy and qPCR)
3. Transfer of patients to Ban Lung hospital for a 7-days clinical follow-up
4. Blood collection followed by CQ administration
5. Parasite clearance and whole blood CQ concentration follow-up during 7 days.
6. Parasitemia follow-up during 2 months with patients staying in Ban Lung during the entire study to make sure no re-infection occurs (Ban Lung is a no-transmission area).
7. Ex vivo drug susceptibility assay of P. vivax isolates and after any recrudescence/relapse, if any.
8. Genotyping analysis of parasites at Day 0 and after any recrudescence/relapse, if any.

Research design

The study will be carried out in Ban Lung district (Rattanakir province, Cambodia) between April 2014 and December 2014. This research site (Rattanakiri) is chosen on the basis of relatively high reports of treatment failures to CQ. In Ban Lung district villages, all P. vivax mono-infected adult patients seeking treatment at community level (VMW and Health centers) will be offered to participate to the study

The sample size calculation was based on addressing the primary objective of identifying a true resistance phenotype to CQ. Therefore a minimum of 50 patients is required and ideally, around 100 patients will increase the probability of detecting resistant parasites.

All eligible participants will be approached by the study staff and information about the objectives of the study will be explained. Informed consent will be obtained from each participant before inclusion.

All P. vivax mono-infected patients identified in the study sites will be included.

Staff involved in this research study will be composed from scientists and technicians from CNM and IPC. Additional collaborators (Reference hospital, Health centers and VMW staff ion Rattanakiri province) will be involved in the project.

Villages in Ban Lung district where P. vivax transmission occur will be selected. Patients seeking treatment from those villages (VMW and Health canters) will be tested for malaria infection by RDT and any non-P. falciparum infected patient will be offered to participate to the study. Falciparum malaria cases will be managed by VMW and Health centers as usually according to Cambodian National guidelines

After obtaining informed consent, the patients will be enrolled in the study and two groups will be constituted:

1. a control group of patients staying in their village and
2. a group transferred to Banlung hospital.

Then, 3 x 5ml-ACD tubes of venous blood will be collected prior to be given CQ to patients.

For the control group, parasitemia will be followed at Day3, D7, D14, D28 and D42 D49, D56 and D60 according to WHO protocol, using fingerprick-collected blood.

For the study group, patients will be followed by fingerprick for parasites clearance and CQ concentration measures every 8h for at least 3 days until complete parasite clearance (determined by two consecutive negative results in microscopy and qPCR). Parasitemia and CQ concentration will be determined daily using fingerprick for 7 days.

To make sure the patients will not be re-infected, they will stay in Ban Lung accommodation for 2 months with every 48h fingerpricks to detect any increase in parasitemia during the study, while the control group will stay in their village where re-infection can occur.

If recrudescence is observed, patients will then be re-admitted in Ban Lung hospital and the same protocol will be performed again.

Ex vivo drug sensitivity assay of the P. vivax isolates will be performed either directly from the blood samples or after cryopreservation. In both case, the assay will involve the invasion of freshly added reticulocytes to the P. vivax isolates.

The reticulocytes used for this work will be obtained from cord blood acquired through the gynecology/obstetric department of Calmette hospital (Pr Kruy Leang Sim), according to the agreement between IPC and Calmette hospital. Cord blood will be supplied regularly to IPC, three times a week, 5 to 7 ml per ACD-tube, 5 tubes per day, if the number of birth allows such sampling. ABO blood group, hemoglobin electrophoresis, G6PD enzyme activity and Duffy status of the blood will be determined before using reticulocytes for P. vivax invasion and culture.

Data will be entered and processed using Microsoft Excel. Parasitemia will be directly correlated to CQ concentration in blood and will allow categorizing the parasites according to the slope of their clearance time and their sensitivity to CQ.

Statistical analysis will be performed when required to detect any significant effects.

ELIGIBILITY:
Inclusion Criteria:

(i) Being aged 15 years or more with competency to give informed consent, (ii) Being positive for P. vivax and mono-infected

Exclusion Criteria:

(i) Being aged 14 years or less (ii) Individuals with illness that affected competency to give informed consent, (iii) Pregnant or lactating women (iv) Having taken antimalarial drugs in the past month

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with P. vivax CQ resistant parasite | 6 months
  Based on parasite clearance time (slow versus fast clearers) and treatments failure (according to the CQ blood concentration)

SECONDARY OUTCOMES:
Number of isolates characterized by whole genome sequencing and multiple Single Nucleotide Polymorphisms Bar Code | 1 year
  P. vivax Isolates will be characterize by SNPs barcode and whole genome sequencing. The final objective is to defined correlations between SNPs detected by whole genome sequencing or bar coding and in vivo and in vitro phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Dysoley Lek, MD, Principal Investigator — National Centre for Parasitology Entomology and Malaria Control; Didier Ménard, PharmD, PhD, Principal Investigator — Institut Pasteur in Cambodia; Jean Popovici, PhD, Principal Investigator — Institut Pasteur in Cambodia
Locations (1):
- Provincial Hospital, Banlung, Ratanakiri, Cambodia

REFERENCES:
- [Derived] Popovici J, Friedrich LR, Kim S, Bin S, Run V, Lek D, Cannon MV, Menard D, Serre D. Genomic Analyses Reveal the Common Occurrence and Complexity of Plasmodium vivax Relapses in Cambodia. mBio. 2018 Jan 23;9(1):e01888-17. doi: 10.1128/mBio.01888-17. PMID 29362233